CLINICAL TRIAL: NCT03717597
Title: A Nonrandomized Evaluation of a Multidimensional Behavioral Intervention for Those at Risk for Alzheimer's Dementia
Brief Title: Nonrandomized Evaluation of a Multidimensional Behavioral Intervention
Acronym: BBLite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1210286
Record Dates: First submitted 2018-05-15; First posted 2018-10-24 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Subjective Cognitive Concerns (SCC)
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: While subjects will be enrolled in multiple groups, all subjects will receive the same intervention and will complete the same study activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will complete an initial assessment within 2 weeks prior to starting the course or during the first class. The course will include 10 sessions conducted on a weekly basis. Following completion of the course, participants will again complete another assessment during the last class or within 2 weeks of course completion. Participants may be invited to complete assessments at 3- and 6-months following course completion.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Subjects will attend a series of 2 hour classes, once a week for 10 weeks. Topics discussed in group sessions will cover compensation strategies (e.g., calendar, goal setting and task lists, functional zones) and brain health behaviors (e.g., exercise, cognitive activity, stress reduction and mindfulness).
  Subjects may be asked to wear an actigraphy monitor (that looks like a wrist watch) and/or heart rate sensor that is designed to collect information regarding physical activity.

SUMMARY:
This intervention is designed to promote enhanced use of compensation strategies including calendar and task list use, and organization systems, as well as increased engagement with brain health activities including physical exercise, cognitive activities, and stress reduction.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and efficacy of a 10-week multi-dimensional intervention for older adults with subjective cognitive concerns (SCC). The goal of this intervention is to enhance compensation skills related to everyday executive and everyday memory functions through training in the systematic use of a calendar system, goal setting and task list system, and organizational strategies within the context of the individual's daily life. This multidimensional intervention program also targets engagement in healthy lifestyle activities (physical exercise, intellectual stimulation, positive emotional functioning) to further promote brain health and functional resilience. Importantly, both treatment components work synergistically as the use of compensation strategies assists in building healthy activities into daily routines (e.g., scheduling exercise into one's calendar and putting it on a task list).

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of subjective cognitive complaints (SCC)
* Age 65+
* English speaking
* Available informant to complete surveys
* Ambulatory

Exclusion Criteria:

* Known neurological condition
* Severe psychiatric illness (e.g., current depression)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Change in compensation use | baseline and 6 months follow up
  Measured using the Everyday Compensation Questionnaire, a 54-item self-report questionnaire that asks participants how often they engage in a variety of activities that help them stay cognitively and physically active.
Change in cognition | baseline and 6 months follow up
  Measured using the Everyday Cognition (ECog) scale, a self-rated questionnaire of cognitively-based everyday abilities. The ECog comprises of 39 items on which the participant's current level of everyday functioning is compared to 10 years earlier. Items are rated on a four-point scale: 1= better or no change compared to 10 years earlier; 4= consistently much worse. Higher scores indicate greater functional limitations.

SECONDARY OUTCOMES:
Beck Depression Inventory | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  Measures depressive symptomatology
Beck Anxiety Inventory | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  measures anxiety symptomatology
List learning task | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  measures learning and memory
Executive function task | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  measures executive function
Psychomotor Speed Task | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  measures psychomotor function
GRIT | baseline, immediately after intervention, and 3 and 6 month follow-up visits
  8-item questionnaire assessing consistency of interest and perseverance of effort on a five-point scale: 1 = not at all like me, 5 = very much like me.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chan, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomaszewski Farias S, Schmitter-Edgecombe M, Weakley A, Harvey D, Denny KG, Barba C, Gravano JT, Giovannetti T, Willis S. Compensation Strategies in Older Adults: Association With Cognition and Everyday Function. Am J Alzheimers Dis Other Demen. 2018 May;33(3):184-191. doi: 10.1177/1533317517753361. Epub 2018 Jan 23. PMID 29357670
- [Background] Farias ST, Lau K, Harvey D, Denny KG, Barba C, Mefford AN. Early Functional Limitations in Cognitively Normal Older Adults Predict Diagnostic Conversion to Mild Cognitive Impairment. J Am Geriatr Soc. 2017 Jun;65(6):1152-1158. doi: 10.1111/jgs.14835. Epub 2017 Mar 17. PMID 28306147
- [Background] Greenaway MC, Duncan NL, Smith GE. The memory support system for mild cognitive impairment: randomized trial of a cognitive rehabilitation intervention. Int J Geriatr Psychiatry. 2013 Apr;28(4):402-9. doi: 10.1002/gps.3838. Epub 2012 Jun 7. PMID 22678947
- [Background] Greenaway MC, Hanna SM, Lepore SW, Smith GE. A behavioral rehabilitation intervention for amnestic mild cognitive impairment. Am J Alzheimers Dis Other Demen. 2008 Oct-Nov;23(5):451-61. doi: 10.1177/1533317508320352. PMID 18955724
- [Background] Lau KM, Parikh M, Harvey DJ, Huang CJ, Farias ST. Early Cognitively Based Functional Limitations Predict Loss of Independence in Instrumental Activities of Daily Living in Older Adults. J Int Neuropsychol Soc. 2015 Oct;21(9):688-98. doi: 10.1017/S1355617715000818. Epub 2015 Sep 22. PMID 26391766